CLINICAL TRIAL: NCT02003183
Title: FDDNP-PET Imaging in Persons at Risk for Chronic Traumatic Encephalopathy
Brief Title: Traumatic Brain Injury and Risk for Chronic Traumatic Encephalopathy
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Gary Small, MD, Principal Investigator, University of California, Los Angeles
Other Study IDs: 11-001077; IND 74944 (Other: FDA)
Record Dates: First submitted 2013-11-05; First posted 2013-12-06 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: CTE; TBI (Traumatic Brain Injury)
Keywords: Chronic Traumatic Encephalopathy; Traumatic Brain Injury; Cognitive Impairment; Positron Emission Tomography; [F-18]FDDNP
MeSH Terms: conditions — Brain Injuries, Traumatic; Chronic Traumatic Encephalopathy; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Samples are being stored
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Suspected CTE: A total of 22 participants with suspected CTE were studied. Each received clinical and neuropsychological assessments, [F-18]FDDNP-PET scans, and magnetic resonance imaging (MRI) scans, or computed tomography scans if they could not tolerate MRI (to assist in PET region of interest identification).
  Interventions: Radiation: [F-18]FDDNP

INTERVENTIONS:
Radiation: [F-18]FDDNP — Each participant was injected with [F-18]FDDNP, a radiolabeled molecular imaging probe, prior to receiving a PET scan.

SUMMARY:
This project was designed to determine brain imaging patterns using 2-(1-{6-[(2-fluorine 18-labeled fluoroethyl)methylamino]-2-naphthyl}ethylidene)malononitrile ([F-18]FDDNP) with positron emission tomography (PET) in participants with suspected Chronic Traumatic Encephalopathy (CTE), a progressive degenerative disease of the brain found in people with a history of repetitive traumatic brain injuries (TBIs), characterized by personality, behavioral, and mood disturbances, cognitive impairment, and sometimes motor symptoms. Currently, CTE can only be definitely diagnosed from neuropathological examination of the brain after autopsy. Developing tools to assist in the detection of this condition in living individuals at risk would facilitate research focusing on discovering potential prevention and treatment strategies.

DETAILED DESCRIPTION:
The project involved clinical and neuropsychological evaluations of participants with histories of TBI and symptoms suggestive of CTE; performing [F-18]FDDNP-PET scans on those participants; determining if patterns of [F-18]FDDNP binding in the brain differ from those of normal controls and Alzheimer's dementia (AD) (available from other studies). Prior research has shown that [F-18]FDDNP-PET produces binding patterns in the brain that indicate high concentrations of tau neurofibrillary tangles (NFTs) and amyloid plaques (Small et al, 2006).

The investigators aimed to test the following hypothesis: [F-18]FDDNP-PET scans will demonstrate cerebral patterns of binding in participants with suspected CTE that differ from cerebral patterns observed in cognitively-intact control participants and participants with AD. The [F-18]FDDNP-PET binding patterns are expected to be consistent with known plaque and tangle deposition patterns from previous neuropathology studies.

[F-18]FDDNP is a PET molecular imaging probe with high in vitro binding affinity to amyloid plaques, NFTs and fibrillar tau deposits as shown with fluorescent microscopy with non-radioactive FDDNP.

In addition to the above hypothesis, neuropathological data from autopsy follow-up (when it becomes available) will be used to determine correlations between regional plaque and tangle deposition patterns observed in neuropathological studies with imaging results from [F-18]FDDNP scans.

Background:

Emerging evidence indicates that repetitive, mild TBI may have long lasting effects following exposure during contact sports or military activities. As a result of recent military conflicts, a high proportion of U.S. veterans have returned from the wars in Iraq and Afghanistan with head injuries resulting from non-penetrating mechanisms.

The syndrome of CTE has been described in previous research performed on contact-sport athletes and military veterans (Omalu et al, 2005, 2006, 2010). In addition, studies of retired professional football players have demonstrated a high rate of dementia, AD, mild cognitive impairment, and depression (Guskiewicz et al, 2005, 2007).

Chronic Traumatic Encephalopathy consists of a characteristic neurobehavioral syndrome manifested by impaired personal and professional functioning, emotional disturbances, depression, alcohol and substance abuse, cognitive impairment, and suicidal behavior. It typically begins after a latency period of several years following single or repeated TBIs. A history of cerebral concussion may or may not be present. The neuroanatomical correlate consists of a tauopathy, the abnormal staining indicative of tau protein deposition in neuronal cell bodies and their axonal and dendritic connections. These representative changes of NFTs and neuritic threads are characteristic of CTE, and distinguish it from other forms of neurodegeneration.

Chronic Traumatic Encephalopathy has a classical distribution that differs than other forms of neurodegeneration (Barrio et al, 2015). The areas of involvement are the temporal and frontal cortices, in addition to the mesencephalon and upper pons, locus coeruleus, and substantia nigra. This distribution, along with the history of multiple exposures to mild TBI, the age distribution, and anatomical patterns further distinguishes this condition from AD and other forms of dementia.

Currently, the only method to diagnose CTE is through post-mortem brain examination, using special immuno-staining techniques for tau protein deposits in NFTs and neuritic threads. The ability to image tau protein collections in vivo in the form of NFTs would provide tremendous benefit for clinical management, treatment, and possibly prevention if a pre-morbid diagnosis could be confirmed. The implications for the sports communities, military organizations, and the general population, all of whom have potential exposure to TBI, are tremendous.

UCLA scientists have developed an in vivo method to measure NFTs, fibrillar tau deposits, and amyloid plaques in the brain. This discovery was led by Dr. Jorge Barrio (Department of Molecular and Medical Pharmacology), Dr. Gary Small (UCLA Division of Geriatric Psychiatry), and others. They sought a way to directly measure the physical evidence of AD - amyloid plaques and tau NFTs - in the living patient. A key to the discovery was the realization that the internal environments of these abnormal proteins were hydrophobic, that is, less friendly to water than to fat. Dr. Jorge Barrio synthesized a new group of compounds that thrived in these hydrophobic environments, and these molecules passed easily from the blood stream to brain tissues.

In initial autopsy studies, the UCLA group found that one of these new compounds (called FDDNP - UCLA Patent Ref. No. 1998-507-1) clearly displayed the well-defined characteristics needed to image these abnormal protein deposits. They then injected a radioactive form of the compound into the veins of living AD patients, and the PET scan accurately measured the concentration and location of the compound in the patient's brain. This allowed them to see for the first time, increased signals coming from living human brains in areas that contained dense collections of the abnormal proteins. .

The chemical marker essentially seeks out and temporarily attaches itself to the abnormal amyloid and tau deposits, thus providing a PET scan signal in the areas of the brain where the proteins are present in high concentrations. In healthy people without AD, these brain regions produce little or no signal. However, in people with the disease, the signal is so strong and accurate that it actually correlates with each individual's degree of memory impairment. The UCLA group has also found that people who are at risk for AD (mild cognitive impairment) have an [F-18]FDDNP signal pattern intermediate between cognitively-intact participants and those with AD, and that participants with a genetic risk for AD show higher [F-18]FDDNP binding (Small et al, 2006, 2009). Therefore, this technology could assist in early detection of the disease so that prevention treatments might be used prior to significant cognitive decline. It will also be useful in detecting and developing treatments for other conditions. Patients with dementias that have different treatment approaches (e.g., frontotemporal) have an an [F-18]FDDNP-PET pattern distinct from AD, as do patients with cognitive impairment associated with prion disease (Kepe et al, 2010).

ELIGIBILITY:
Inclusion Criteria:

1. Agreement to participate in study;
2. A history of TBI resulting from, but not limited to, any of the following: contact sports, accidents, violence, or military combat;
3. Age 18 or older;
4. No significant cerebrovascular disease;
5. Adequate visual and auditory acuity to allow neuropsychological testing;
6. Screening laboratory tests without significant abnormalities that might interfere with the study.

Exclusion Criteria:

1. Preexisting major neurological or other physical illness that could confound results (e.g., multiple sclerosis, diabetes, cancer);
2. History of myocardial infarction within the previous year or unstable cardiac disease.
3. Uncontrolled hypertension (systolic blood pressure > 170 or diastolic blood pressure > 100),
4. History of significant liver disease, clinically significant pulmonary disease, diabetes, or cancer.
5. Such current major psychiatric disorders as mania within the previous two years.
6. Participants taking drugs that are known to affect [F-18]FDDNP-PET binding (e.g., ibuprofen, naproxen) were asked to stop taking medication one week prior to PET scan or excluded from the study.
7. Use of any investigational drugs within the previous month, depending on drug half-life.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Military personnel and retired football players were exclusively men, whereas the comparative groups (AD, cognitively healthy controls) had a substantial proportion of women. Military personnel were significantly younger than the other three groups. Four of the seven military personnel were cognitively normal, and three had mild cognitive impairment. While the difference in education levels among participant groups did not reach statistical significance, pairwise comparisons indicated that military personnel had significantly lower education levels than both players and cognitively healthy individuals. Military personnel and players had significantly higher levels of depression and anxiety than did the comparison groups.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary W Small, M.D., Principal Investigator — UCLA Division of Geriatric Psychiatry
Locations (1):
- UCLA Division of Geriatric Psychiatry, Semel Institute, Los Angeles, California, United States

REFERENCES:
- [Background] Omalu BI, DeKosky ST, Hamilton RL, Minster RL, Kamboh MI, Shakir AM, Wecht CH. Chronic traumatic encephalopathy in a national football league player: part II. Neurosurgery. 2006 Nov;59(5):1086-92; discussion 1092-3. doi: 10.1227/01.NEU.0000245601.69451.27. PMID 17143242
- [Background] Omalu BI, DeKosky ST, Minster RL, Kamboh MI, Hamilton RL, Wecht CH. Chronic traumatic encephalopathy in a National Football League player. Neurosurgery. 2005 Jul;57(1):128-34; discussion 128-34. doi: 10.1227/01.neu.0000163407.92769.ed. PMID 15987548
- [Background] Guskiewicz KM, Marshall SW, Bailes J, McCrea M, Harding HP Jr, Matthews A, Mihalik JR, Cantu RC. Recurrent concussion and risk of depression in retired professional football players. Med Sci Sports Exerc. 2007 Jun;39(6):903-9. doi: 10.1249/mss.0b013e3180383da5. PMID 17545878
- [Background] Guskiewicz KM, Marshall SW, Bailes J, McCrea M, Cantu RC, Randolph C, Jordan BD. Association between recurrent concussion and late-life cognitive impairment in retired professional football players. Neurosurgery. 2005 Oct;57(4):719-26; discussion 719-26. doi: 10.1093/neurosurgery/57.4.719. PMID 16239884
- [Background] Omalu BI, Bailes J, Hammers JL, Fitzsimmons RP. Chronic traumatic encephalopathy, suicides and parasuicides in professional American athletes: the role of the forensic pathologist. Am J Forensic Med Pathol. 2010 Jun;31(2):130-2. doi: 10.1097/PAF.0b013e3181ca7f35. PMID 20032774
- [Background] Small GW, Kepe V, Ercoli LM, Siddarth P, Bookheimer SY, Miller KJ, Lavretsky H, Burggren AC, Cole GM, Vinters HV, Thompson PM, Huang SC, Satyamurthy N, Phelps ME, Barrio JR. PET of brain amyloid and tau in mild cognitive impairment. N Engl J Med. 2006 Dec 21;355(25):2652-63. doi: 10.1056/NEJMoa054625. PMID 17182990
- [Background] Small GW, Siddarth P, Burggren AC, Kepe V, Ercoli LM, Miller KJ, Lavretsky H, Thompson PM, Cole GM, Huang SC, Phelps ME, Bookheimer SY, Barrio JR. Influence of cognitive status, age, and APOE-4 genetic risk on brain FDDNP positron-emission tomography imaging in persons without dementia. Arch Gen Psychiatry. 2009 Jan;66(1):81-7. doi: 10.1001/archgenpsychiatry.2008.516. PMID 19124691
- [Background] Kepe V, Ghetti B, Farlow MR, Bresjanac M, Miller K, Huang SC, Wong KP, Murrell JR, Piccardo P, Epperson F, Repovs G, Smid LM, Petric A, Siddarth P, Liu J, Satyamurthy N, Small GW, Barrio JR. PET of brain prion protein amyloid in Gerstmann-Straussler-Scheinker disease. Brain Pathol. 2010 Mar;20(2):419-30. doi: 10.1111/j.1750-3639.2009.00306.x. Epub 2009 Jun 9. PMID 19725833
- [Result] Small GW, Kepe V, Siddarth P, Ercoli LM, Merrill DA, Donoghue N, Bookheimer SY, Martinez J, Omalu B, Bailes J, Barrio JR. PET scanning of brain tau in retired national football league players: preliminary findings. Am J Geriatr Psychiatry. 2013 Feb;21(2):138-44. doi: 10.1016/j.jagp.2012.11.019. Epub 2013 Jan 22. PMID 23343487
- [Result] Barrio JR, Small GW, Wong KP, Huang SC, Liu J, Merrill DA, Giza CC, Fitzsimmons RP, Omalu B, Bailes J, Kepe V. In vivo characterization of chronic traumatic encephalopathy using [F-18]FDDNP PET brain imaging. Proc Natl Acad Sci U S A. 2015 Apr 21;112(16):E2039-47. doi: 10.1073/pnas.1409952112. Epub 2015 Apr 6. PMID 25848027
- [Result] Chen ST, Siddarth P, Merrill DA, Martinez J, Emerson ND, Liu J, Wong KP, Satyamurthy N, Giza CC, Huang SC, Fitzsimmons RP, Bailes J, Omalu B, Barrio JR, Small GW. FDDNP-PET Tau Brain Protein Binding Patterns in Military Personnel with Suspected Chronic Traumatic Encephalopathy1. J Alzheimers Dis. 2018;65(1):79-88. doi: 10.3233/JAD-171152. PMID 30040711
- [Result] Omalu B, Small GW, Bailes J, Ercoli LM, Merrill DA, Wong KP, Huang SC, Satyamurthy N, Hammers JL, Lee J, Fitzsimmons RP, Barrio JR. Postmortem Autopsy-Confirmation of Antemortem [F-18]FDDNP-PET Scans in a Football Player With Chronic Traumatic Encephalopathy. Neurosurgery. 2018 Feb 1;82(2):237-246. doi: 10.1093/neuros/nyx536. PMID 29136240

RESULTS

PARTICIPANT FLOW:
Groups:
- Military Personnel: Military personnel with suspected chronic traumatic encephalopathy (CTE), each with a history of head trauma and cognitive or mood symptoms.
- Players: Retired football players with suspected CTE, each with a history of head trauma and cognitive or mood symptoms.
Period: Overall Study
Arm/Group | Military Personnel | Players
Started | 7 | 17
Completed | 7 | 15
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants had suspected CTE because of a history of traumatic brain injury and cognitive and/or mood symptoms. Of the 24 participants, 2 were lost to follow up and not included in the data analysis.
Groups:
- Military Personnel: Military personnel with a history of head trauma and cognitive or mood symptoms.
- Players: Retired football players with a history of head trauma and cognitive or mood symptoms.
- Total: Total of all reporting groups
Arm/Group | Military Personnel | Players | Total
Number analyzed (Participants) | 7 | 15 | 22
Age, Continuous [Mean (Full Range); unit: years] | 45 [33 to 57] | 54 [40 to 86] | 49 [33 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 15 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 4 | 10 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Distribution Volume Ratio (DVR)
Description: The outcome measure is a ratio of the volume (in milliliters) of 2-(1-{6-[(2-fluorine 18-labeled fluoroethyl)methylamino]-2-naphthyl}ethylidene)malononitrile ([F-18]FDDNP) bound within the region of interest (ROI) divided by the amount of [F-18]FDDNP in the cerebellum (reference region). Higher ratios are indicative of higher levels of tau and amyloid proteins within the ROI. The unit of measure is called the Distribution Volume Ratio (DVR).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Distribution Volume Ratio (DVR)
Arm/Group | Military Personnel | Players
Number analyzed (Participants) | 7 | 15
Distribution Volume Ratio (DVR)
  Amygdala | 1.30 (0.09) | 1.39 (.10)
  Midbrain | 1.26 (0.14) | 1.34 (0.07)
  Hypothalamus | 1.32 (.13) | 1.42 (.08)
  Thalamus | 1.37 (.14) | 1.51 (.10)
  Pons | 1.27 (.14) | 1.31 (.07)
  Striatum (caudate nucleus and putamen) | 1.33 (.10) | 1.53 (.10)
Statistical Analysis 1: Comparison: Military Personnel vs Players; This analysis applies to the Amygdala; Test type: Superiority; p < 0.02, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = .09, Standard Deviation .1

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Military Personnel | Players
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/15
Other Adverse Events (participants affected / at risk) | 0/7 | 0/15

LIMITATIONS AND CAVEATS:
Although the participants groups were matched for important variables, these results need interpretation with caution given the relatively small sample sizes. Differences in cerebrovascular health and other variables also could influence the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-03): https://cdn.clinicaltrials.gov/large-docs/83/NCT02003183/Prot_SAP_000.pdf